CLINICAL TRIAL: NCT05159245
Title: The Finnish National Study to Facilitate Patient Access to Targeted Anti-cancer Drugs to Determine the Efficacy in Treatment of Advanced Cancers With a Known Molecular Profile
Brief Title: The Finnish National Study to Facilitate Patient Access to Targeted Anti-cancer Drugs
Acronym: FINPROVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Katriina Jalkanen, Chief Physician, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FINPROVE
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Advanced Cancer; Solid Tumor; Haematological Malignancy
Keywords: DRUP study
MeSH Terms: conditions — Hematologic Neoplasms | interventions — alectinib; cobimetinib; HhAntag691; entrectinib; atezolizumab; Vemurafenib; regorafenib; apalutamide; abemaciclib; tepotinib; dabrafenib; trametinib; pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (15):
- Alectinib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by alectinib.
  Interventions: Drug: Alectinib
- Cobimetinib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by cobimetinib.
  Interventions: Drug: Cobimetinib
- Vismodegib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by vismodegib.
  Interventions: Drug: Vismodegib
- Trastuzumab+Pertuzumab (Experimental): For patients with a molecular tumor profile that can potentially be targeted by trastuzumab+pertuzuma combination.
  Interventions: Drug: Trastuzumab+Pertuzumab
- Entrectinib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by entrectinib.
  Interventions: Drug: Entrectinib
- Atezolizumab (Experimental): For patients with a molecular tumor profile that can potentially be targeted by atezolizumab.
  Interventions: Drug: Atezolizumab
- Vemurafenib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by vemurafenib.
  Interventions: Drug: Vemurafenib
- Regorafenib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by regorafenib.
  Interventions: Drug: Regorafenib
- Apalutamide (Experimental): For patients with a molecular tumor profile that can potentially be targeted by apalutamide.
  Interventions: Drug: Apalutamide
- Abemaciclib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by abemaciclib.
  Interventions: Drug: Abemaciclib
- Tepotinib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by tepotinib.
  Interventions: Drug: Tepotinib
- Dabrafenib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by dabrafenib.
  Interventions: Drug: Dabrafenib
- Trametinib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by trametinib.
  Interventions: Drug: Trametinib
- Dabrafenib+Trametinib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by dabrafenib+trametinib combination.
  Interventions: Drug: Dabrafenib+Trametinib
- Pemigatinib (Experimental): For patients with a molecular tumor profile that can potentially be targeted by pemigatinib.
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Alectinib — ALK
  Other Names: Alecensa
  Arms: Alectinib
Drug: Cobimetinib — MEK1, MEK2
  Other Names: Cotellic
  Arms: Cobimetinib
Drug: Vismodegib — Hedgehog
  Other Names: Erivedge
  Arms: Vismodegib
Drug: Trastuzumab+Pertuzumab — HER2
  Other Names: Phesgo
  Arms: Trastuzumab+Pertuzumab
Drug: Entrectinib — NTRK/ ROS1, ALK
  Other Names: Rozlytrek
  Arms: Entrectinib
Drug: Atezolizumab — PD-L1
  Other Names: Tecentriq
  Arms: Atezolizumab
Drug: Vemurafenib — BRAF V600
  Other Names: Zelboraf
  Arms: Vemurafenib
Drug: Regorafenib — KIT/BRAF, RET
  Other Names: Stivarga
  Arms: Regorafenib
Drug: Apalutamide — AR
  Other Names: Erleada
  Arms: Apalutamide
Drug: Abemaciclib — CDK4/6
  Other Names: Verzenio
  Arms: Abemaciclib
Drug: Tepotinib — MET ex14
  Other Names: Tepmetko
  Arms: Tepotinib
Drug: Dabrafenib — RAF
  Other Names: Tafinlar
  Arms: Dabrafenib
Drug: Trametinib — MEK1, MEK2
  Other Names: Mekinist
  Arms: Trametinib
Drug: Dabrafenib+Trametinib — RAF, MEK1, MEK2
  Other Names: Tafinlanr+Mekinist
  Arms: Dabrafenib+Trametinib
Drug: Pemigatinib — FGFR2
  Other Names: Pemazyre
  Arms: Pemigatinib

SUMMARY:
This is a prospective non-randomized national clinical phase 2 trial that aims to determine the efficacy and toxicity of targeted anticancer drugs or combinations that are approved or under review by EMA, FDA or PMDA and are used for treatment of patients with advanced cancer with a potentially actionable variant as revealed by a genomic, RNA-molecular or protein expression test.

DETAILED DESCRIPTION:
This is a prospective non-randomized clinical trial that aims to determine the efficacy and toxicity of targeted anticancer drugs or combinations that are approved or under review by EMA, FDA or PMDA and are used for treatment of patients with advanced cancer with a potentially actionable variant as revealed by a genomic, RNA-molecular or protein expression test. The study also aims to facilitate patient access to approved targeted therapies that are contributed to the program by collaborating pharmaceutical companies and to perform next generation sequencing and further deeper analysis on tumor biopsies and/or liquid biopsies for biomarker analyses and resistance mechanisms. Eligible patients have an advanced cancer for which standard treatment options no longer exist and acceptable performance status and organ function. A tumour DNA, RNA or protein expression analysis is required and the results must identify at least one potentially actionable molecular variant as defined in the protocol. Molecular profiling will be utilized to determine an appropriate drug(s) from among those available in the protocol. Drug selection will be guided by a list of potential profiles, the molecular tumor board and databases of identified targets for review and approval of the recommended treatment. The protocol-specified treatment will be administered to the patient once any drug- and disease specific eligibility criteria and overall study criteria are met. Data for standard efficacy outcomes including tumor response, progression-free and overall survival as well as duration of treatment will be collected for all patients receiving treatment within the trial. In addition, treatment related toxicity will be collected according to CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age >18 years) patient with a histologically-confirmed locally advanced or metastatic cancer who is no longer benefitting from standard anti-cancer treatment or for whom no such treatment is available or indicated.
2. ECOG performance status 0-2
3. Patients must have acceptable organ function as defined below. However, specific inclusion/exclusion criteria specified in the drug-specific study manual will take precedence:

   1. Absolute neutrophil count ≥ 1.5 x 109/l
   2. Hemoglobin > 8.0 mmol/l, without blood transfusion within 7 days
   3. Platelets > 75 x 109/l (not applicable for hematological patients)
   4. Total bilirubin < 1.5 x ULN
   5. AST and ALT < 3 x institutional ULN (or < 5 x ULN in patients with known hepatic metastases)
   6. Serum creatinine ≤ 1.5 × ULN or calculated or measured creatinine clearance ≥ 40 mL/min/1.73 m2
4. Patients must have objectively evaluable or measurable disease (by physical or radiographic examination, according to RECIST v1.1, Lugano, IWG and ELN-AML, IMWG, RANO, GCIG, iRESIST or PCWG3.
5. Results must be available from a tumor molecular profiling. Eligible tests may include any of the following technologies: fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR), comparative genomic hybridization (CGH), next generation sequencing (NGS) or immunohistochemistry (IHC). The test may have been performed on the primary tumor or a metastatic lesion, in a diagnostic laboratory or within the context of another commercial platform (eg Foundation Medicine), and must reveal a potentially actionable variant.
6. Patients must have a tumor profile for which treatment with one of the approved (or under revision for approval) targeted anti-cancer drugs included in this study has potential clinical benefit based on preclinical data or clinical information.
7. A new (obtained ≤6 months before inclusion after which no further anti-cancer therapy is allowed) fresh frozen and FFPE tumor biopsy specimen or liquid biopsy for extensive biomarker testing is mandatory before the start of treatment with a targeted agent included in the protocol.
8. Ability to understand and the willingness to sign a written informed consent document and comply to the protocol.
9. For orally administered drugs, the patient must be able to swallow and tolerate oral medication and must have no known malabsorption syndrome.
10. Because of the risks of drug treatment to the developing fetus, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation, and for four months following completion of study therapy. Male patients should avoid impregnating a female partner. Male patients, even if surgically sterilized, (i.e. post-vasectomy) must agree to one of the following: practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or completely abstain from sexual intercourse.

Exclusion Criteria:

1. Ongoing toxicity > grade 2, other than alopecia or > grade 1 neuropathy.
2. Patient is receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement). Required wash out period prior to starting study treatment is at least two weeks. An exception is made for:

   1. Patients suffering from CRPC are allowed to continue androgen deprivation therapy.
   2. Medications that are prescribed for supportive care but may potentially have an anti-cancer effect (e.g., megestrol acetate, bisphosphonates). These medications must have been started ≥ 1 week prior to enrollment on this study.
3. Received colony-stimulating factors (eg, G-CSF, GM-CSF or recombinant EPO) within 14 days prior to the first dose of study intervention
4. Patient is pregnant or nursing.
5. Patients with known active progressive brain metastases. Patients with previously treated brain metastases are eligible, provided that the patient is clinically stable and off steroids for at least 4 weeks prior to study initiation. GMB patients apply additional exclusion criteria.
6. Patients with clinically significant preexisting cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure are not eligible.
7. Patients with clinically significant preexisting cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure are not eligible.
8. Patients with known left ventricular ejection fraction (LVEF) < 45% are not eligible
9. Patients with stroke (including TIA) or acute myocardial infarction within 3 months before the first dose of study treatment are not eligible
10. Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements including, but not limited to: ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness/social situations.

For each drug included in this protocol, specific inclusion and exclusion criteria (based on the Package Insert or manufacturers recommendations) may also apply. Drug-specific inclusion and exclusion criteria will take precedence over the inclusion/exclusion criteria listed above.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 16 weeks
  Disease control rate at 16 weeks after treatment initiation (defined as patients by CR, PR, SD)

SECONDARY OUTCOMES:
Duration of treatment | 5 years
  Time on drug
Adverse Events | 5 years
  Treatment-related grade ≥3 and serious adverse events
Overall response | 5 years
  Best overall response (defined as patients by CR, PR, SD)
PFS | 5 years
  Progression free survival
OS | 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Katriina Jalkanen, MD, PhD, Principal Investigator — Helsinki University Hospital Comprehensive Cancer Centre
Locations (5):
- Finland (5):
  - Turku University Hospital Cancer Centre, Turku, Southwest Finland
  - Helsinki University Hospital Comprehensive Cancer Center, Helsinki, Uusimaa
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital OYS Cancer Center, Oulu
  - Tampere University Hospital Department of Oncology, Tampere

IPD SHARING:
Plan to Share IPD: Yes
Investigators plan to share the clinical study report.
Supporting Information: CSR
Time Frame: 2026-2027
Access Criteria: Will be made available through European regulatory CTIS programme.